CLINICAL TRIAL: NCT04431908
Title: Validation of a Rapid Quantitative Test for Loss of Smell in COVID-19 Subjects
Status: Completed | Type: Observational
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Other Study IDs: 2000028259
Record Dates: First submitted 2020-06-12; First posted 2020-06-16 (Actual); Results first posted 2021-06-02 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: COVID-19
Keywords: olfactory device; COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Outpatients (Drive Thru): Patients receiving testing through a drive thru location.
  Interventions: Device: olfactory device
- High Risk Asymptomatics: Asymptomatic patients (residents) in a high risk location.
  Interventions: Device: olfactory device

INTERVENTIONS:
Device: olfactory device — A quantitative non-biased olfactory device intended for the rapid identification of SARS-CoV-2 infected subjects (as identified by PCR).

SUMMARY:
The purpose of this study is to evaluate the performance of a non-invasive olfactory device as a rapid indicator of COVID-19 in positive subjects.

DETAILED DESCRIPTION:
The major hypothesis is that a quantitative and unbiased smell test will be a useful tool to identify COVID-19 positive individuals.

The study will address what fraction of outpatients truly have a loss-of-smell (including a partial loss) and is expected to outperform the current question that is used to identify COVID-19 related anosmia "Do you have a new loss of smell or taste?" (yes/no) in terms of sensitivity and specificity.

The study will address if high-risk asymptomatic people whom are SARS-CoV-2 positive have a partial (or perhaps transitory) loss of smell.

The primary objective of this study is to validate the utility (sensitivity, specificity and accuracy) of a quantitative non-biased olfactory device for the rapid identification of SARS-CoV-2 infected subjects (as identified by PCR). The performance of the device will also be compared to the standard CDC patient query for 'new loss of smell or taste'.

The secondary objective is to test if SARS-CoV-2 positive 'asymptomatic' COVID-19 subjects may actually present with a mild or transitory defect in smell (hyposmia), which is revealed through our quantitative olfactory smell test.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Have a corresponding PCR test for SARS-CoV-2 on the same day.

Exclusion Criteria:

* Adults unable to consent
* Individuals who are not yet adults (infants, children, teenagers)
* Pregnant women
* Individuals with allergic to fragrances
* History of surgery on the nose or paranasal sinuses
* Asthmatics
* Patients with known neurocognitive disorders: dementia, Alzheimer's disease, Parkinson's disease
* Adults with Acute or Chronic rhinosinusitis (They will be asked if they have a 'stuffy or runny nose'; they may be included in some tests, but their analysis would be segregated as they may be false positives due to allergies or a common cold or flu)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The population will be either individuals receiving drive-thru COVID-19 testing or residents of a nursing facility receiving tests.
Sampling Method: Non-Probability Sample
Enrollment: 1320 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2020-10-15 (Actual); Study Completion 2020-11-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: R Peter Manes, MD, FACS, Principal Investigator — Associate Professor of Surgery (Otolaryngology)
Locations (1):
- Yale New Haven Hospital, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Patel RA, Torabi SJ, Kasle DA, Manes RP. Five-item odorant test as an indicator of COVID-19 infection in a general population. Am J Otolaryngol. 2022 Mar-Apr;43(2):103376. doi: 10.1016/j.amjoto.2022.103376. Epub 2022 Jan 29. PMID 35151176

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We did end up testing more individuals than expected due to increased ability
Groups:
- High Risk Asymptomatics: Asymptomatic patients (health care workers) in a high risk location.
  olfactory device: A quantitative non-biased olfactory device intended for the rapid identification of SARS-CoV-2 infected subjects (as identified by PCR).
Period: Overall Study
Arm/Group | Outpatients (Drive Thru) | High Risk Asymptomatics
Started | 1042 | 278
Completed | 1042 | 278
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Outpatients (Drive Thru) | High Risk Asymptomatics | Total
Number analyzed (Participants) | 1042 | 278 | 1320
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 878 | 251 | 1129
  >=65 years | 164 | 27 | 191
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 615 | 200 | 815
  Male | 427 | 78 | 505
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Race and Ethnicity data were not collected for the purposes of this study.
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Race and Ethnicity data were not collected for the purposes of this study.
Region of Enrollment [Number; unit: participants]
  United States | 1042 | 278 | 1320

OUTCOME MEASURES:

1. Primary Outcome: Sensitivity, Specificity and Accuracy
Description: The subject's score on using the olfactory device will be compared to the PCR results (SARS-CoV-2 negative or positive) on COVID19 outpatients. As the smell test has a variable scale (0-5) the ideal cutoff will be determined to maximize these factors:
  * Sensitivity (Represents True Positives Divided by True Positives plus False Negatives)
  * Specificity (Represents True Negatives Divided by True Negatives plus False Positives)
  * Accuracy (Represents Sensitivity x Prevalence + Specificity x (1-Prevalence) True Positives are patients who got 3 or less correct answers on the smell test and had a positive PCR COVID test.
  True Negatives are patients who got 4 or 5 correct responses on the smell test and had a negative PCR COVID test.
  False Positives are patients who got 3 or less correct responses on the smell test and had a negative PCR COVID test.
  False Negatives are patients who got 4 or 5 correct responses on the smell test and had a positive PCR COVID test.
Time Frame: 24 hours
Population: Only participants in the drive thru were analyzed for this outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | Outpatients (Drive Thru)
Number analyzed (Participants) | 1042
Participants
  True Negative | 889
  False Positive | 106
  False Negative | 27
  True Positive | 20
Statistical Analysis 1: Comparison: Outpatients (Drive Thru); Test type: Other — Sensitivity, specificity and accuracy was measured utilizing the true and false positives, as well as the true and false negatives. For a subject to have a true positive, the subject must have had a positive PCR test for COVID-19 as well as scored 0, 1 or 2 correct answers on the smell test. For a subject to have a true negative, the subject must have had a negative PCR test for COVID-19 as well as scored 3, 4 or 5 correct answers on the smell test; Specificity = 89.35
Statistical Analysis 2: Comparison: Outpatients (Drive Thru); Test type: Other — [test comment as in outcome 1, analysis 1]; Sensitivity = 42.55
Statistical Analysis 3: Comparison: Outpatients (Drive Thru); Test type: Other — [test comment as in outcome 1, analysis 1]; Accuracy = 87.24

2. Secondary Outcome: Repeatability
Description: Repeatability will also be examined in a test-retest score conducted within 24 hours with a second device in which the sequence of the odorants is altered.
Time Frame: 48 hours
Population: It was not feasible to get return visits as intended in the proposed protocol and therefore these data were not collected.
Arm/Group | Outpatients (Drive Thru) | High Risk Asymptomatics
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Asymptomatic Sensitivity, Specificity and Accuracy
Description: We will determine if 'asymptomatic' SARS-CoV-2 positive subjects experience a partial loss of smell (hyposmia) and if so determine the fraction of subjects in which this occurs. We will evaluate sensitivity, specificity and accuracy.
  Sensitivity (Represents True Positives Divided by True Positives plus False Negatives)
  * Specificity (Represents True Negatives Divided by True Negatives plus False Positives)
  * Accuracy (Represents Sensitivity x Prevalence + Specificity x (1-Prevalence) True Positives are patients who got 3 or less correct answers on the smell test and had a positive PCR COVID test.
  True Negatives are patients who got 4 or 5 correct responses on the smell test and had a negative PCR COVID test.
  False Positives are patients who got 3 or less correct responses on the smell test and had a negative PCR COVID test.
  False Negatives are patients who got 4 or 5 correct responses on the smell test and had a positive PCR COVID test.
Time Frame: 24 hours
Population: Only asymptomatic patients were analyzed for this outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | High Risk Asymptomatics
Number analyzed (Participants) | 278
Participants
  True Negative | 244
  False Positive | 31
  False Negative | 27
  True Positive | 1
Statistical Analysis 1: Comparison: High Risk Asymptomatics; Test type: Other — [test comment as in outcome 1, analysis 1]; Specificity = 88.73
Statistical Analysis 2: Comparison: High Risk Asymptomatics; Test type: Other — [test comment as in outcome 1, analysis 1]; Sensitivity = 33.33
Statistical Analysis 3: Comparison: High Risk Asymptomatics; Test type: Other — [test comment as in outcome 1, analysis 1]; Accuracy = 88.13

ADVERSE EVENTS:
Time Frame: An average of 30 minutes after administration of the smell test
Description: Serious and Other Adverse Event definitions do not differ from those of ClinicalTrials.gov
Arm/Group | Outpatients (Drive Thru) | High Risk Asymptomatics
All-Cause Mortality (participants affected / at risk) | 0/1042 | 0/278
Serious Adverse Events (participants affected / at risk) | 0/1042 | 0/278
Other Adverse Events (participants affected / at risk) | 0/1042 | 0/278

LIMITATIONS AND CAVEATS:
It is possible that the PCR COVID test results were incorrect, as these tests are not 100% accurate.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-01): https://cdn.clinicaltrials.gov/large-docs/08/NCT04431908/Prot_SAP_000.pdf